CLINICAL TRIAL: NCT04982796
Title: Psilocybin-Enhanced Psychotherapy for Methamphetamine Use Disorder
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Portland VA Research Foundation, Inc (Other)
Collaborators: Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Amphetamine-Related Disorders
Keywords: methamphetamine, stimulant, psilocybin, psychedelic, psychotherapy
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical interviewers will be blinded to condition and study timepoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin-enhanced psychotherapy (Experimental): Psilocybin will be administered twice (25mg & 30mg two weeks apart) in addition to a 6-week psychotherapy protocol while admitted to a residential rehabilitation treatment program.
  Interventions: Drug: Psilocybin; Behavioral: Treatment-as-usual
- Treatment-as-Usual (Other): Treatment-as-usual while admitted to a residential rehabilitation treatment program.
  Interventions: Behavioral: Treatment-as-usual

INTERVENTIONS:
Drug: Psilocybin — See description of psilocybin-enhanced psychotherapy arm.
  Arms: Psilocybin-enhanced psychotherapy
Behavioral: Treatment-as-usual — See description of treatment-as-usual arm.

SUMMARY:
This is a proof-of-concept randomized clinical trial of psilocybin-enhanced psychotherapy versus treatment-as-usual among individuals being treated for methamphetamine use disorder.

DETAILED DESCRIPTION:
The trial will take place with individuals admitted to a residential rehabilitation treatment program. The treatment protocol will consist of 4 preparatory therapy visits, 2 psilocybin sessions (25-30mg), and 8 total integration therapy visits. Primary aims assess acceptability, feasibility, and safety with a primary endpoint at the conclusion of the study intervention. An additional aim assesses preliminary efficacy for methamphetamine use disorder and overall functioning at follow-up assessments 60 and 180 days after discharge from the residential treatment program.

ELIGIBILITY:
Inclusion Criteria:

* United States military Veteran
* Moderate to severe methamphetamine use disorder using the DSM-V diagnostic criteria
* Desire to cease or reduce methamphetamine use

Exclusion Criteria:

* Have uncontrolled hypertension or clinically significant cardiovascular disease
* History of seizure disorder in adulthood
* CNS metastases or symptomatic central nervous system (CNS) infection
* Poorly controlled diabetes mellitus
* Taking certain medications that may interact with psilocybin
* History of any primary persistent psychotic disorder, including schizophrenia, schizoaffective disorder, bipolar disorder with psychosis, major depressive disorder with psychosis, or schizophreniform disorder
* History of bipolar I disorder
* Current eating disorder with active purging
* History of hallucinogen use disorder
* Pregnant or breast feeding

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability | End of 6-week intervention; approximately 42 days
  We will use a 7-point Likert scale to measure each participant's perceived benefit and perceived harm of the intervention.
Proportion of patients who complete the intervention and follow-up | End of 6-week intervention to 180 days post-discharge follow-up; approximately 180 days
  We will observe the proportion of patients who complete the intervention and follow-up to determine feasibility.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 180 day post-discharge follow-up; approximately 222 days post-enrollment
  Number of Participants Who Experienced Treatment-related Adverse Events as defined by the FDA (21 Code of Federal Regulations [CFR] 312.32(a)). Adverse events assessed at every study visit by clinical observation and patient interview.
Methamphetamine Use, self-report | 60 days post-discharge follow-up; approximately 102 days post-enrollment
  Using the Timeline Follow-Back procedure, average number of days per week used methamphetamine over the past four weeks.
Methamphetamine Use, self-report | 180 days post-discharge follow-up; approximately 222 days post-enrollment
  Using the Timeline Follow-Back procedure, average number of days per week used methamphetamine over the past four weeks.
Methamphetamine Use, urine | 60 days post-discharge follow-up; approximately 102 days post-enrollment
  Urine drug screen
Methamphetamine Use, urine | 180 days post-discharge follow-up; approximately 222 days post-enrollment
  Urine drug screen
Change from baseline in Sheehan Disability Scale (SDS) at end-of-intervention | approximately 42 days post-enrollment
  Sheehan Disability Scale total score, a measure of clinician-rated functional impairment. SDS scores range from 0 (not impaired) to 30 (highly impaired).
Change from baseline in Sheehan Disability Scale at 60 day post-discharge follow-up | approximately 102 days post-enrollment
  Sheehan Disability Scale total score, a measure of clinician-rated functional impairment
Change from baseline in Sheehan Disability Scale at 180 day post-discharge follow-up | approximately 222 days post-enrollment
  Sheehan Disability Scale total score, a measure of clinician-rated functional impairment

OTHER OUTCOMES:
Change from baseline in Stimulant Craving at end-of-intervention | approximately 42 days post-enrollment
  Stimulant Craving Questionnaire-Brief
Change from baseline in Stimulant Craving at 60 day post-discharge follow-up | approximately 102 days post-enrollment
  Stimulant Craving Questionnaire-Brief
Change from baseline in Stimulant Craving at 180 day post-discharge follow-up | approximately 222 days post-enrollment
  Stimulant Craving Questionnaire-Brief
Change from baseline in Depression Symptoms at end-of-intervention | approximately 42 days post-enrollment
  Beck Depression Inventory-II
Change from baseline in Depression Symptoms at 60 day post-discharge follow-up | approximately 102 days post-enrollment
  Beck Depression Inventory-II
Change from baseline in Depression Symptoms at 180 day post-discharge follow-up | approximately 222 days post-enrollment
  Beck Depression Inventory-II
Change from baseline in PTSD Symptoms at end-of-intervention | approximately 42 days post-enrollment
  PTSD Checklist for Diagnostic and Statistical Manual (DSM)-5
Change from baseline in PTSD Symptoms at 60 day post-discharge follow-up | approximately 102 days post-enrollment
  PTSD Checklist for DSM-5
Change from baseline in PTSD Symptoms at 180 day post-discharge follow-up | approximately 222 days post-enrollment
  PTSD Checklist for DSM-5
Change from baseline in Anxiety Symptoms at end-of-intervention | approximately 42 days post-enrollment
  Measured by Generalized Anxiety Disorder-7 (GAD-7). Scores range from 0 (minimal anxiety) to 21 (severe anxiety).
Change from baseline in Anxiety Symptoms at 60 day post-discharge follow-up | approximately 102 days post-enrollment
  Generalized Anxiety Disorder-7
Change from baseline in Anxiety Symptoms at 180 day post-discharge follow-up | approximately 222 days post-enrollment
  Generalized Anxiety Disorder-7
Change from baseline in Attachment Insecurity at end-of-intervention | approximately 42 days post-enrollment
  Experiences in Close Relationships-Short form
Change from baseline in Attachment Insecurity at 60 day post-discharge follow-up | approximately 102 days post-enrollment
  Experiences in Close Relationships-Short form
Change from baseline in Attachment Insecurity at 180 day post-discharge follow-up | approximately 222 days post-enrollment
  Experiences in Close Relationships-Short form
Change from baseline in Immune Markers at end-of-intervention | approximately 42 days post-enrollment
  C-Reactive Protein, Interleukin (IL)-6, Tumor Necrosis Factor (TNF)-a, IL-8, IL-10, IL-1β, CCL2, CCL3
Change from baseline in Heart Rate Variability at end-of-intervention | approximately 42 days post-enrollment
  heart rate variability, 7 minutes, resting

CONTACTS AND LOCATIONS:
Overall Officials: Chris Stauffer, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Portland VA Health Care System, Vancouver, Washington, United States

IPD SHARING:
Plan to Share IPD: No